CLINICAL TRIAL: NCT06904118
Title: Clinical Efficacy of Novel Titanium Oxide Nanoparticle Enriched Bleaching Gel on Tooth Whitening and Hypersensitivity: A Randamized Clinical Trial.
Brief Title: Clinical Efficacy of Novel Titanium Oxide Nanoparticle Enriched Bleaching Gel
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pakistan Institute of Medical Sciences (Other Government)
Responsible Party: Principal Investigator, Afsheen Mansoor, Principal Investigator, Pakistan Institute of Medical Sciences
Allocation: Non-Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SOD/ ERB/2023/31-01
Record Dates: First submitted 2025-03-25; First posted 2025-04-01 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Tooth Discoloration; Tooth Sensitivity
Keywords: Biowaste,; Hypersensitivity; Silky Corn Hair Fiber; Titanium oxide nanoparticles (TiO2 Nps); whitening
MeSH Terms: conditions — Tooth Discoloration; Dentin Sensitivity; Hypersensitivity

STUDY DESIGN:
Intervention Model Description: Interventional Study Model: Parallel Assignment
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Triple (Participant, Care Provider, Outcomes Assessor) In this triple-blind trial, participants, care provider and outcome assessor were unaware of the study groups
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group-A (Experimental): Experimental: Group A (Nano-reinforced Hydrtogen peroxide ) Nano-reinforced hydrogen peroxide bleaching gel
  Interventions: Drug: Nano-reinforced Novel Hydrogen peroxide gel
- Group-B (Experimental): Group-B (Conventional Hydrogen peroxide) Conventional Hydrogen peroxide gel without nanoparticles
  Interventions: Drug: Conventional Hydrogen peroxide gel without nanoparicles

INTERVENTIONS:
Drug: Nano-reinforced Novel Hydrogen peroxide gel — Group A (Novel Nano-enriched Hydrogen peroxide bleaching gel with Silky Corn hair fiber derived- titania nanoparticles)
  Arms: Group-A
Drug: Conventional Hydrogen peroxide gel without nanoparicles — Drug: Hydrogen peroxide without nanoparicles Group B ( Conventional Hydrogen peroxide gel without nanoparticles)
  Arms: Group-B

SUMMARY:
The goal of this clinical trial is to learn the effect of Nano-fortified Bleaching on whitening and sensitivity of teeth.The main questions it aims to answer are:

Does Nano-fortified Bleaching gel is more effective in enhancing the whitening in comparison to conventional bleaching gel ? Does Nano-fortified Bleaching gel is more effective in declining the sensitivity in comparison to conventional bleaching gel ?

Participants will be divided into 2 groups i.e Group A where Nano-fortified Bleaching agent will be employed and Group B where Conventional Bleaching agent without nanoparticles will be used. One application of bleaching for thirty minutes will be carried out . Tooth sensitivity will be measured by VAS Scale having "No Pain" at one-end and "Worst Pain" at opposite-end .Color change will be measured with spectrophotometer.

DETAILED DESCRIPTION:
This triple blinded randomized clinical trial will be performed where Participants without any caries, restorations or periodontal disease in anterior teeth having shade A3 or darker will be included in this trial. Those having poor oral hygiene; caries, restorations, periodontal disease, root canal treatment, fractures, gingival recessions, cervical lesions, bruxism, severe internal discoloration, dental prosthesis, cracks and spontaneous TS, in anterior teeth will be excluded. Consecutive non probability sampling technique will be used where total participants (n=60) will be randomly allocated into two groups 'A' and 'B' (n= 30). After informed consent, bleaching protocol will be carried out in both the groups 'A' and 'B'with conventional and novel bleaching gel. The color change (ΔE) and post bleaching hypersensitivity scores will be recorded by Visual analogue scale (VAS). In group A; Nano-fortified Novel TiHP gel (Titanium Dioxide nanoparticles and 35 % Hydrogen Peroxide ) will be used for the participants of Group-A and Conventional bleaching gel (35 % Hydrogen Peroxide) will be utilized for participants of Group-B. The color change (ΔE) will be investigated via spectrophotometer and VAS score will be calculated by participants who will be instructed to rate their hypersensitivity scores after 1st session, 2nd session, 3rd session and post-bleaching after 1 week and 1 month

ELIGIBILITY:
Inclusion Criteria:Patients enrolled in the current trial ranged between 20- 40 years old with good general and oral health. Participants selected without any caries, restorations or periodontal disease in anterior teeth. The selected participants possessed maxillary incisors having shade A3 or darker after checking with Vita Classical Shade Guide

Exclusion Criteria:The patients having poor oral hygiene; caries, restorations, periodontal disease, root canal treatment, fractures, gingival recessions, cervical lesions, bruxism, severe internal discoloration, dental prosthesis, cracks and spontaneous TS, in anterior teeth shall be excluded from this study. Moreover, pregnant, lactating women, smokers, patients taking medications, those having fixed orthodontic appliances and undergone tooth whitening will be also excluded

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2023-06-13 (Actual); Primary Completion 2023-12-27 (Actual); Study Completion 2023-12-27 (Actual)

PRIMARY OUTCOMES:
Post-bleaching sensitivity | 3 months
  Pain scores assessed by Visual Analogue Scale (VAS) score after 4hr, 24hrs, 48hrs, 72hrs, 96hrs. The minimum score is O (None) and the maximum score is 10 (Severe)

SECONDARY OUTCOMES:
Post-bleaching whitening | 3 months
  Color change shall be measured with spectrophotometer; and calculated through formula; ΔE = [(ΔL*)2 + (Δa*)2 + (Δb*)2 ] 1/2 with different readings taken by two calibrated evaluators.

CONTACTS AND LOCATIONS:
Overall Officials: Afsheen Mansoor, PhD, Principal Investigator — School of Dentistry, Shaheed Zulfiqar Ali Bhutto Medical University, Islamabad.
Locations (1):
- School of Dentistry, Pakistan Institute of Medical Sciences, Islamabad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Coppla FM, Rezende M, de Paula E, Farago PV, Loguercio AD, Kossatz S, Reis A. Combination of Acetaminophen/Codeine Analgesics Does Not Avoid Bleaching-Induced Tooth Sensitivity: A Randomized, Triple-Blind Two-Center Clinical Trial. Oper Dent. 2018 Mar/Apr;43(2):E53-E63. doi: 10.2341/17-092-C. PMID 29504880
- See also: Coppla, F. M., Rezende, M., de Paula, E., Farago, P. V., Loguercio, A. D., Kossatz, S., & Reis, A. (2018). Combination of Acetaminophen/Codeine Analgesics Does Not Avoid Bleaching-Induced Tooth Sensitivity: A Randomized, Triple-Blind Two-Center Clinical — https://pubmed.ncbi.nlm.nih.gov/29504880/